CLINICAL TRIAL: NCT04393675
Title: Clinical Pharmacology of LT5001 Drug Product in Hemodialysis Patients With Uremic Pruritus to Assess the Safety, Local Tolerance and Pharmacokinetics
Brief Title: Study to Investigate the Safety of LT5001 Drug Product for Uremic Pruritus in Hemodialysis Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in the clinical development plan
Sponsor: Lumosa Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT5001-101
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Uremic Pruritus
Keywords: uremic pruritus; Hemodialysis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LT5001 (Active Comparator): Administered twice daily (maximum 6 g per time, morning and evening respectively)
  Interventions: Drug: LT5001
- Placebo (Placebo Comparator): Administered twice daily (maximum 6 g per time, morning and evening respectively)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LT5001 — LT5001 is administered twice daily.
  Arms: LT5001
Drug: Placebo — LT5001 is administered twice daily.
  Arms: Placebo

SUMMARY:
A Randomized, Double Blind, Placebo-Controlled study to assess the Safety, Local Tolerance, and Pharmacokinetics of LT5001 drug product in Hemodialysis Patients with Uremic Pruritus

DETAILED DESCRIPTION:
In Part A, patient participation is expected to last up to 63 days, including a 28-day screening period(consisting of a 7-day diary run-in to build baseline itch NRS) and a 36-day on study period (consisting of 56 total doses from Day 1 to Day 29, and a 7 day follow-up/EOS visit at Day 36).

In Part B, patient participation is expected to last up to 85 days, including a 28-day screening period (consisting of a 7-day diary run-in to build baseline itch NRS) and a 57-day on study treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 20 to 75 years of age, inclusive, at the time of signing informed consent.
2. Patient must have been receiving in-center hemodialysis for ≥ 3 months and currently on a schedule of 3 times per week.
3. Patient must have had at least 2 urea reduction ratio (URR) measurements ≥ 65%, at least 2 single-pool Kt/V measurements ≥ 1.2, or 1 single-pool Kt/V measurement ≥ 1.2 and 1 URR measurement ≥ 65% on different dialysis days within the last 3 month period prior to the Screening Visit.
4. Body weight ≥ 40 kg (not to exceed 115 kg) and BMI ≥ 18.0 and ≤ 31.0 kg/m2 at screening and Day 1 (after hemodialysis).
5. History of pruritus > 4 weeks of duration
6. Females with childbearing potential (defined as women ≤50 years of age with a history of amenorrhea for <12 months prior to study entry) must agree to use effective methods of contraception from screening through the last dose of study drug.
7. Males who are sexually active and whose partners are females of childbearing potential must agree to use condoms from screening through 90 days, whichever is longer, after administration of the last dose of study drug, and their partners must be willing to use a highly effective method of contraception from screening through 90 days after administration of the last dose of study drug.
8. Males must agree to not donate sperm from screening through 90 days, whichever is longer, after administration of the last dose of study drug.
9. Patient must have completed at least 6 days of Worst Itching Intensity NRS worksheets in the 7-day Diary run-in period and have a mean Worst Itching Intensity NRS score > 4 prior to randomization.
10. Patients must be able to complete questionnaires, understand the study procedures, and communicate effectively with the study personnel.

Exclusion Criteria:

1. History of alcohol abuse, illicit drug use, physical dependence to any opioid or narcotic, or any history of drug abuse or addiction within 6 months of screening.
2. History of major surgery or trauma within 12 weeks of screening in the judgement of the investigator, or surgery planned during the study.
3. Has received ultraviolet B treatment, opioid antagonists (eg, naloxone, naltrexone), or opioid mixed agonist-antagonist (eg, nalbuphine) within 30 days prior to the Screening Visit or anticipated to receive such treatment during the study.
4. Has had a significant alteration in dialysis regimen within 2 weeks of the Screening Visit or anticipated to be receiving nocturnal dialysis, home hemodialysis treatment, or kidney transplant during the study.
5. Has any known history of allergic reaction to opioids.
6. History of latest positive serology test for HBV (HBsAg) or HCV (anti-HCV) within 1 year prior randomization consistent with current infection. Confirmatory tests will be allowed at the discretion of the investigator to rule out false positives.
7. Has any known history of HIV.
8. Positive pregnancy test or is lactating.
9. Has required peritoneal dialysis.
10. Alanine aminotransferase and/or aspartate aminotransferase concentration > 2 x the ULN, or total bilirubin > 1.8 x ULN, or hemoglobin concentration < 9 g/dL at the Screening Visit.
11. Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half-lives (if known) of the investigational drug's PK, PD, or biological activity (if known), whichever is longer, prior to first dose of study drug in this study or is currently participating in another clinical study.
12. Has received a vaccination within 3 days prior to administration of the first dose of study drug.
13. Has pruritus probably or definitely attributed to a cause other than renal disease or its complications such as atopic dermatitis, chronic urticarial, or hepatic pruritus caused by chronic liver disease.
14. Presence of skin infection (as defined by the investigator) on the area to be treated.
15. Any other condition or prior therapy that, in the investigator's opinion, would make the patient unsuitable for the study, or unable or unwilling to comply with the study procedures
16. Involved in the planning or conduct of this study.
17. Unwilling or unlikely to comply with the requirements of the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: June Kuo, Study Director — Lumosa Therapeutics
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated after completion of Part A (18 participants). Part B was planned but not initiated.
Pre-assignment Details: Participants underwent a 7-day run-in period prior to Part A. Only participants meeting eligibility criteria after the run-in period were enrolled into Part A. No participants entered Part B, as Part B was not initiated.
Groups:
- LT5001: LT5001 group
- Placebo: Placebo as control
Period: Part A
Arm/Group | LT5001 | Placebo
Started | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0
Period: Part B (Not Initiated)
Arm/Group | LT5001 | Placebo
Started (did not initiated) | 0 | 0 (did not initiated)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 12 participant in the LT5001 group; 6 in the placebo group
Groups:
- LT5001; Placebo: Administered twice daily
- Total: Total of all reporting groups
Arm/Group | LT5001 | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (5.9) | 53.8 (12.7) | 56.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 12 | 6 | 18
weight [Mean (Standard Deviation); unit: kilogram] | 58.3 (13.9) | 67.0 (16.7) | 61.2 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Events With AE by Severity
Description: The number of reported AE events by severity
Time Frame: Week 4
Population: Safety population: include all patients who receive at least 1 dose of LT5001 drug product or placebo
Measure: Number; unit: events
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
events
  Any TEAE by severity -Mild | 6 | 2
  Any TEAE by severity -Moderate | 0 | 0
  Any TEAE by severity -Severe | 1 | 0

2. Primary Outcome: Number of Patients With AE by Severity
Description: Adverse events (AEs) were collected and categorized by severity (mild, moderate, or severe) according to standard clinical criteria. The outcome measure is defined as the number of patients who experienced at least one adverse event of each severity level during the study period.
Time Frame: Week 4
Population: include all patients who receive at least 1 dose of LT5001 drug product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
Participants
  Mild | 6 | 1
  Moderate | 0 | 0
  Severe | 1 | 0

3. Primary Outcome: The Number of Patients With AE by Causality
Description: Adverse events were assessed for their causal relationship to the study treatment by the investigator and categorized as related or not related. The outcome measure is defined as the number of patients who experienced at least one adverse event in each causality category during the study period.
Time Frame: 4 weeks
Population: Include all patients who receive at least 1 dose of LT5001 drug product or placebo
Measure: Number; unit: participants
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
participants
  unrelated | 5 | 1
  unlikely | 0 | 0
  Possibly | 1 | 0
  Probably | 0 | 0
  Definitely | 0 | 0

4. Primary Outcome: Number of AE Event by Causality
Description: The number of reported events by causality
Time Frame: week 4
Population: include all patients who receive at least 1 dose of LT5001 drug product or placebo
Measure: Number; unit: events
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
events
  unrelated | 6 | 2
  unlikely | 0 | 0
  possibly | 1 | 0
  probably | 0 | 0
  definitely | 0 | 0

5. Secondary Outcome: Systemic Ctrough Exposure of LT5001 in Hemodialysis Patients.
Description: The systemic trough (Ctrough) concentration of LT5001 was measured in hemodialysis patients at specified time points prior to the next scheduled dose using validated bioanalytical methods. The outcome measure is defined as the plasma concentration of LT5001 immediately before each dosing interval.
Time Frame: Week 4
Population: include patients who have received at least 1 dose of LT5001 drug product and have at least 1 measured concentration of LT5001 drug product at a scheduled PK time point after dosing.
Measure: Mean (Standard Deviation); unit: ng/ml of LT5001 in blood
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
ng/ml of LT5001 in blood | NA (NA) — below the limit of quantification (BLQ) | NA (NA) — below the limit of quantification (BLQ)

6. Secondary Outcome: Change in Mean Worst Itching Intensity From Baseline to the End of Week 4 Using NRS.
Description: The intensity of itch will be measured using the Numerical Rating Scale (NRS), a standardized scale for assessing the worst itching over the past 24 hours. The scale ranges from 0 to 10, where 0 represents no itching and 10 represents the worst itching imaginable. Higher scores indicate worse itch severity. The outcome measure is defined as the change in mean worst itching intensity from baseline to the end of Week 4.
Time Frame: Week 4
Population: include all randomized patients who received at least 1 dose of LT5001 drug product or placebo
Measure: Mean (Standard Deviation); unit: score on the Numerical Rating Scale (NRS
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
score on the Numerical Rating Scale (NRS | -1.8 (2.1) | -2.3 (2.4)

7. Secondary Outcome: Proportion of Patients With Changes in Numerical Rating Scale (>=2 Points, >=3 Points, >=4 Points) From Baseline
Description: The Numerical Rating Scale (NRS) is an 11-point scale used to assess itch intensity, where scores range from 0 to 10, with 0 indicating no pain and 10 indicating the worst itch imaginable. A decrease in NRS score represents an improvement in itch severity. This outcome measures the proportion of patients who achieved a reduction of at least 2 points, 3 points, or 4 points from baseline in NRS score at Week 4.
Time Frame: Week 4
Population: include all randomized patients who received at least 1 dose of LT5001 drug product or placebo
Measure: Number; unit: participants
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
participants
  >=2 points >=2 points >=2 points >=2 points >= 2 points | 5 | 3
  >= 3 points | 2 | 2
  >= 4 points | 1 | 2

8. Secondary Outcome: Improvement in Itch-related Quality of Life as Assessed by the Change From Baseline in 5-D Pruritus Scale at the End of Week 4.
Description: The 5-D Pruritus Scale (5-D Itch Scale) is a multidimensional questionnaire assessing itching across five key domains: Duration, Degree, Direction, Disability, and Distribution, to comprehensively evaluate the impact of itch on daily life. The scale ranges from 5 to 25, with 5 representing no itch and 25 representing severe itch. Each domain is scored from 1 (lowest) to 5 (highest). Higher scores indicate worse itch and poorer itch-related quality of life, whereas lower scores indicate better quality of life. The outcome measure is defined as the change from baseline in 5-D Pruritus Scale total score at the end of Week 4, with improvement reflected by a decrease in total score.
Time Frame: Week 4
Population: include all randomized patients who received at least 1 dose of LT5001 drug product or placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
score on a scale | -3.2 (2.9) | -3.8 (1.6)

9. Secondary Outcome: Improvement in Itch-related Quality of Life as Assessed by the Change From Baseline in Total Skindex-10 Scale Score at the End of Week 4.
Description: The Skindex-10 Scale is a multidimensional questionnaire assessing itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. Each of the 10 items is scored from 0 to 6, resulting in a total score ranging from 0 to 60, where 0 represents never bothered/no impact and 60 represents always bothered/severe impact. Higher scores indicate worst itch-related quality of life, whereas lower scores indicate better quality of life. The outcome measure is defined as the change from baseline in total Skindex-10 Scale Score at the end of Week 4, with improvement reflected by a decrease in total score.
Time Frame: Week 4
Population: include all randomized patients who received at least 1 dose of LT5001 drug product or placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LT5001 | Placebo
Number analyzed (Participants) | 12 | 6
score on a scale | -15.1 (11.2) | -22.2 (3.6)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 5 weeks
Arm/Group | LT5001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/6
Other Adverse Events (participants affected / at risk) | 7/12 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LT5001 (N=12) | Placebo (N=6)
vitreous haemorrhage (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LT5001 (N=12) | Placebo (N=6)
skin rash (Skin and subcutaneous tissue disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Toxic goitre (Endocrine disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04393675/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04393675/SAP_001.pdf